CLINICAL TRIAL: NCT06529146
Title: Real-World Data Study Assessing the Efficacy of Troriluzole-Treated Subjects With Spinocerebellar Ataxia (SCA) Compared to a Matched External SCA Control Using Natural History Cohort Data
Brief Title: Real-World Data Study of Troriluzole-Treated Patients With Spinocerebellar Ataxia (SCA) Compared to a Matched Natural History Control
Status: Active, not recruiting | Type: Observational
Sponsor: Biohaven Therapeutics Ltd. (Industry)
Responsible Party: Sponsor
Organization: Biohaven Pharmaceuticals, Inc. (Industry)
Other Study IDs: BHV4157-206-RWE
Record Dates: First submitted 2024-07-26; First posted 2024-07-31 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Spinocerebellar Ataxias
Keywords: propensity score match; natural history; disease registry; SCA; f-SARA
MeSH Terms: conditions — Spinocerebellar Ataxias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Troriluzole-treated SCA subjects: The BHV4157-206 study is a Phase III, multicenter, randomized, double-blind, 2-arm, placebo-controlled parallel-group study designed to assess the safety, tolerability, and efficacy of troriluzole in a population of patients with SCA. Subjects were randomized to receive placebo (QD) or troriluzole (200 mg QD). BHV4157-206 consisted of a randomization phase and an OLE phase. Subjects in the trorilzuole-treated cohort are from study BHV4157-206, were originally randomized to troriluzole, and extended an opportunity to continue treatment in an open-label extenstion (OLE) phase. All subjects had the opportunity to complete 3-years of treatment.
  Interventions: Drug: BHV-4157
- SCA Natural History Comparator: The natural history comparison group includes SCA subjects from the CRC-SCA and EUROSCA natural history studies. The CRC-SCA study includes individuals with SCA 1, 2, 3, 6, 7, 8, and 10, with the time period of data collection spanning 2010 to present. Patients taking riluzole or troriluzole in the CRC-SCA study were not included in this analysis. The EUROSCA study included individuals with SCA genotypes 1, 2, 3, and 6, with the time period of data collection spanning 2005-2009. The natural history protocols were finalized prior to our conduct of the present analysis, as each was designed for independent research purposes.

INTERVENTIONS:
Drug: BHV-4157 — BHV-4157 (troriluzole) 200 mg QD
  Groups: Troriluzole-treated SCA subjects

SUMMARY:
The purpose of this study is to leverage two sources of real-world data (RWD) to assess the effectiveness of troriluzole after three years of treatment in patients with SCA by comparison to an external control of untreated patients who were followed in a natural history cohort.

Real world evidence of effectiveness will be assessed from the RWD sources to examine the treatment effects of toriluzole in SCA out to 3 years. Progression rates of SCA differ by genotype and long-term follow-up is needed to assess for potential efficacy in this rare disease.

DETAILED DESCRIPTION:
This study comprises multiple sources of RWD including: 1) the Clinical Research Consortium for the Study of Cerebellar Ataxia (CRC-SCA/US SCA Natural History cohort; 2) the European Integrated Project on Spinocerebellar Ataxias (EUROSCA/European SCA Natural History Cohort); and 3) the 3 year OLE data from troriluzole treated subjects in Study BHV4157-206 (NCT03701399). Each participant of the study will have their efficacy and/or safety data collected as pre-specified in the original protocols from the RWD sources.

The effectiveness of troriluzole in SCA after 3 years of treatment from the long-term, open-label extension from Study BHV4157-206 will be compared to external control subjects collected from CRC-SCA (US SCA Natural History cohort) and EUROSCA (European SCA Natural History Cohort). A propensity score matching (PSM) analysis will be utilized to create equipoise across groups being examined in the analysis.

The primary outcome will be change from baseline in the modified functional Scale for the Assessment and Rating of Ataxia (f-SARA). Another endpoint examined will be a newly developed and validated composite endpoint for SCA, the Spinocerebellar Ataxia Composite Score (SCACOMS).

ELIGIBILITY:
Key Inclusion Criteria for troriluzole-treated participants (BHV4157-206):

* Between the ages of 18-75
* Genetic confirmation of the following specific hereditary ataxias: SCA1, SCA2, SCA3, SCA6, SCA7, SCA8, and SCA10
* Screening f-SARA total score of ≥3 and score of ≥1 on gait item of the f-SARA.
* Ability to ambulate 8 meters without human assistance (canes and other devices were allowed)
* Subjects initially randomized to troriluzole

Key Inclusion Criteria for participants selected from the natural history studies:

* Between ages of 18-75
* CRC-SCA: either a genetic confirmation or a diagnosis of SCA 1, 2, 3, 6, 7, 8, and 10 in themselves or a family member; EUROSCA: genetic confirmation of SCA genotypes 1, 2, 3 and 6.

Key Exclusion Criteria for troriluzole-treated participants (BHV4157-206 study):

* Screening f-SARA score of 4 on any item of the f-SARA
* Any other medical condition that could predominantly explain or contribute significantly to the subjects' symptoms of ataxia or that could confound assessment of ataxia symptoms

Key Exclusion Criteria for participants selected from the natural history studies:

• Treatment with troriluzole

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study involves the analysis of data collected among three research settings: 1) European registry of SCA patients (2005-2008) (NCT02440763 ); 2) US registry of SCA patients (2010-present) (NCT01060371); 3) Subjects originally randomized to troriluzole in BHV4157-206 with 3-years of treatment data (NCT03701399).
Sampling Method: Non-Probability Sample
Enrollment: 909 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2024-09-06 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the total score of the modified functional Scale for the Assessment and Rating of Ataxia (f-SARA) at Year 3 in troriluzole-treated subjects is compared to natural history subjects from CRC-SCA | Up to 3 years of treatment
  To compare the effectiveness of troriluzole in treating SCA, as measure by the modified functional Scale for the Assessment and Rating of Ataxia (f-SARA), in subjects randomized to treatment with troriluzole relative to natural history controls from the natural history dataset after 3 years of treatment. The f-SARA is a scale with a range of 0 to 16, where an increase in the total score indicates a worsening of symptoms.

SECONDARY OUTCOMES:
Change from baseline in the f-SARA at Year 2 in troriluzole-treated subjects is compared to the change from baseline in the mapped f-SARA at Year 2 in natural history subjects from CRC-SCA | Up to 2 years of treatment
  The f-SARA is a scale with a range of 0 to 16, where an increase in the total score indicates a worsening of symptoms.
Change from baseline in the f-SARA at Year 1 in troriluzole-treated subjects is compared to the change from baseline in the mapped f-SARA at Year 1 in natural history subjects from CRC-SCA | Up to 1 year of treatment
  The f-SARA is a scale with a range of 0 to 16, where an increase in the total score indicates a worsening of symptoms.
Change from baseline in the f-SARA at Year 3 in troriluzole-treated subjects is compared to the change from baseline in the mapped f-SARA at Year 3 in natural history subjects from EUROSCA | Up to 3 years of treatment
  The f-SARA is a scale with a range of 0 to 16, where an increase in the total score indicates a worsening of symptoms.
Change from baseline in the f-SARA at Year 2 in troriluzole-treated subjects is compared to the change from baseline in the mapped f-SARA at Year 2 in natural history subjects from EUROSCA | Up to 2 years of treatment
  The f-SARA is a scale with a range of 0 to 16, where an increase in the total score indicates a worsening of symptoms.
Change from baseline in the f-SARA at Year 1 in troriluzole-treated subjects is compared to the change from baseline in the mapped f-SARA at Year 1 in natural history subjects from EUROSCA | Up to 1 year of treatment
  The f-SARA is a scale with a range of 0 to 16, where an increase in the total score indicates a worsening of symptoms.
Change from baseline in the f-SARA at Year 3 in troriluzole-treated subjects is compared to the change from baseline in the mapped f-SARA at Year 3 in pooled (CRC-SCA and EUROSCA) natural history subjects | Up to 3 years of treatment
  The f-SARA is a scale with a range of 0 to 16, where an increase in the total score indicates a worsening of symptoms.
Change from baseline in the f-SARA at Year 2 in troriluzole-treated subjects is compared to the change from baseline in the mapped f-SARA at Year 2 in in pooled (CRC-SCA and EUROSCA) natural history subjects | Up to 2 years of treatment
  The f-SARA is a scale with a range of 0 to 16, where an increase in the total score indicates a worsening of symptoms.
Change from baseline in the f-SARA at Year 1 in troriluzole-treated subjects is compared to the change from baseline in the mapped f-SARA at Year 1 in pooled (CRC-SCA and EUROSCA) natural history subjects | Up to 1 year of treatment
  The f-SARA is a scale with a range of 0 to 16, where an increase in the total score indicates a worsening of symptoms.
Change from baseline in Spinocerebellar Ataxia Composite Score (SCACOMS) at Year 3 in troriluzole-treated subjects is compared to that of in CRC-SCA natural history subjects | Up to 3 years of treatment
  The SCACOMS (SCA Composite Scale) is a newly developed and validated endpoint for SCA, derived from an analysis of two SCA natural history studies (CRC-SCA and EUROSCA). The score range of SCACOMS is 0-50, where an increase in the total score indicates a worsening of symptoms.
Change from baseline in SCACOMS at Year 2 in troriluzole-treated subjects is compared to that of in CRC-SCA natural history subjects | Up to 2 years of treatment
  The SCACOMS (SCA Composite Scale) is a newly developed and validated endpoint for SCA, derived from an analysis of two SCA natural history studies (CRC-SCA and EUROSCA). The score range of SCACOMS is 0-50, where an increase in the total score indicates a worsening of symptoms.
Change from baseline in SCACOMS at Year 1 in troriluzole-treated subjects is compared to that of in CRC-SCA natural history subjects | Up to 1 year of treatment
  The SCACOMS (SCA Composite Scale) is a newly developed and validated endpoint for SCA, derived from an analysis of two SCA natural history studies (CRC-SCA and EUROSCA). The score range of SCACOMS is 0-50, where an increase in the total score indicates a worsening of symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Biohaven, New Haven, Connecticut, United States